CLINICAL TRIAL: NCT04259255
Title: Radicava® (Edaravone) Findings in Biomarkers From ALS (REFINE-ALS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tanabe Pharma America, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REFINE-ALS
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: biomarkers; edaravone; Radicava®; Radicava ORS®; motor neuron disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Edaravone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Edaravone (Radicava®/Radicava ORS®): During an estimated 12-month period, eligible participants who are prescribed Edaravone within the approved indication will be invited to participate in the study.
  Interventions: Drug: Edaravone (Radicava®/Radicava ORS®)

INTERVENTIONS:
Drug: Edaravone (Radicava®/Radicava ORS®) — Participants will be followed from enrollment up to 24 weeks after treatment initiation (6 treatment cycles - 28 days per cycle, corresponding to a treatment period of approximately 24 weeks) or premature study discontinuation.
  Biomarker testing and clinical assessments will be performed at baseline (at enrollment or before the start of cycle 1), and at cycles 1, 3, and 6. Dosing is 60 mg daily by intravenous infusion for 14 days for the initial treatment cycle, followed by daily dosing on 10 out of 14 days in subsequent treatment cycles.
  Other Names: Radicava®; Radicava ORS®

SUMMARY:
REFINE-ALS is a prospective, observational, longitudinal, multicenter study designed to identify biomarkers to serve as quantifiable biological non-clinical measures of Edaravone effects in ALS. Epigenetic and protein biomarkers will also be investigated.

DETAILED DESCRIPTION:
Treatment will be prescribed by HCPs in accordance with their clinical judgement and the prescribing information for Edaravone. The decision to prescribe Edaravone to the participants should be made separately from the decision to enroll then in the study. There will be no randomized assignments to treatment and no restrictions on the use of commercially available medications (but those participating in an experimental study, even if taking Edaravone, will be excluded). No experimental treatment is evaluated in this study. The intervention is limited to the collection of blood and urine samples for biomarker testing.

During the estimated study period, eligible patients who are prescribed Edaravone within the approved indication will be invited to participate in the study. An initial screening/baseline visit will be scheduled for participants who are considered for study participation.

Participants in this study will be followed from enrollment up to 24 weeks after treatment initiation (6 treatment cycles [each cycle consisting of 28 days], corresponding to a treatment period of approximately 24 weeks) or premature study discontinuation. Throughout the study period, the investigators will record participant baseline and follow-up information and perform clinical and biomarker assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years or older at enrollment
* Sporadic or familial ALS diagnosed as possible, probable, probable-laboratory supported or definite as defined by the World Federation of Neurology revised El Escorial criteria
* Decision made to prescribe Edaravone prior to screening
* Participant will likely be able to obtain commercial Edaravone and likely to complete 6 cycles of treatment, per site investigator estimation
* Participant either naïve to Edaravone or who did not receive any Edaravone does within 1 month prior to screening
* Signed informed consent by the subject, or a witness if a subject cannot read or write or is physically unable to talk or write, obtained before any study-related activities are undertaken

Exclusion Criteria:

* Participant with a contraindication to Edaravone
* Participant is participating in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in participants who have sporadic or familial amyotrophic lateral sclerosis (ALS) as defined by revised El Escorial criteria. Participants must provide written informed consent prior to screening. At screening, eligible patient must be at least 18 years old with a decision made to prescribe Edaravone prior to consenting. Participants who are either Edaravone naïve or who did not receive any Edaravone dose within one month of consenting are eligible for inclusion given they meet all other protocol requirements.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of 8-F2 isoprostanes as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for 8-F2 isoprostanes.
Change in levels of 3-nitrotyrosine (3-NT) as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for 3-NT.
Change in levels of 8-hydroxy-2'-deoxyguanosine (8-OHdG) as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples 8-OHdG.
Change in levels of urate as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for urate.
Change in levels of matrix metalloproteinase-9 (MMP-9) as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for MMP-9.
Change in levels of urinary neutrophin receptor p75 as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for urinary neutrophin receptor p75.
Change in levels of neurofilaments (Nf) (Heavy and Light) as a potential biomarker of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for neurofilaments (Nf) (Heavy and Light).
Change in levels of creatinine as a potential biomarkers of oxidative stress, inflammation or neurodegeneration. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Collection of blood and/or urine samples for creatinine.

SECONDARY OUTCOMES:
Change from baseline in the ALSFRS-R (ALS Functional Rating Scale .Revised) Score | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  The ALSFRS-R is a quickly administered ordinal rating scale (ratings 0-4) used to determine participants' assessment of their capability and independence in 12 functional activities.
Change from baseline in the King's Clinical Staging. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  The King's clinical staging is based on the number of body regions affected by ALS and the presence of respiratory or nutritional failure.
Change from baseline in the ALSAQ-40 (ALS Assessment Questionnaire). | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  The ALSAQ-40 is a questionnaire that consists of 40 questions/items with 5 discrete scales: physical mobility, activities of daily living and independence, eating and drinking, communication, emotional reactions.
Change from baseline in the Appel ALS Score. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  The Appel ALS score consists of five sub-scores: bulbar, respiratory, muscle strength, and lower extremity and upper extremity function.
Change from baseline in slow vital capacity. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  The vital capacity (VC) (percent of predicted normal) will be determined, using the upright slow VC method.
Change from baseline in hand-held dynamometry. | Cycles 1, 3, and 6 of each Edaravone cycle (each cycle is 28 days).
  Hand-held dynamometry (HHD) will be used as a quantitative measure of muscle strength for this study.

CONTACTS AND LOCATIONS:
Overall Officials: James Berry, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (20):
- United States (19):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCLA Als Clinic, Los Angeles, California
  - UC Davis Health, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida, Jacksonville -Neurology Research Department, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mercy Health, Grand Rapids, Michigan
  - Neurology Associates, P.C., Lincoln, Nebraska
  - Las Vegas Clinic, Las Vegas, Nevada
  - OhioHealth, Columbus, Ohio
  - Jefferson Weinberg ALS Center, Philadelphia, Pennsylvania
  - Temple University Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- SunnyBrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry J, Brooks B, Genge A, Heiman-Patterson T, Appel S, Benatar M, Bowser R, Cudkowicz M, Gooch C, Shefner J, Westra J, Agnese W, Merrill C, Nelson S, Apple S. Radicava/Edaravone Findings in Biomarkers From Amyotrophic Lateral Sclerosis (REFINE-ALS): Protocol and Study Design. Neurol Clin Pract. 2021 Aug;11(4):e472-e479. doi: 10.1212/CPJ.0000000000000968. PMID 34476128